CLINICAL TRIAL: NCT02364050
Title: Prospective Data Collection of Elderly Patients (≥ 65 Years) With Diffuse Large B-cell Lymphoma (DLBCL) Receiving at the Time of Diagnosis Multidimensional Geriatric Assessment (VGM)
Brief Title: Prospective Data Collection of Elderly Patients With DLBCL Receiving at the Time of Diagnosis VGM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_Elderly Project
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly patients with DLBCL: Elderly patients (Age ≥ 65 years) with large B-cell lymphoma classified FIT or UNFIT or FRAIL by Multidimensional Geriatric Assessment (MGA)

SUMMARY:
Prospective data collection of a consecutive series of elderly patients with large B-cell lymphoma newly diagnosed, receiving before the start of treatment Multidimensional Geriatric Assessment (VGM) through the use of Activity of Daily Living (ADL), Instrumental Activity of Daily Living (IADL) and Cumulative Illness Rating Scale for Geriatrics (CIRS-G).

DETAILED DESCRIPTION:
Prospective data collection of a consecutive series of elderly patients with large B-cell lymphoma newly diagnosed, receiving before the start of treatment Multidimensional Geriatric Assessment (VGM) through the use of Activity of Daily Living (ADL), Instrumental Activity of Daily Living (IADL) and Cumulative Illness Rating Scale for Geriatrics (CIRS-G) to be defined in 3 categories:

* elderly FIT (ADL 6; IADL 8; 0 score= 3-4, < 5 score=2)
* elderly UNIFIT (ADL 5; IADL 6-7; 0 score= 3-4, 5-8 score=2; ≥ 80 fit)
* elderly FRAIL (ADL ≤ 4; IADL ≤ 5; 1 score= 3-4, > 8 score=2; ≥ 80 unfit)

ELIGIBILITY:
Inclusion Criteria:

* Patient with Large B-cell Lymphoma
* Age ≥ 65 years
* informed Consent

Exclusion Criteria:

* Violation of inclusion criteria
* Abscence of data considered essential for the study
* Withdrawal of Consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with large B-cell lymphoma classified FIT or UNFIT or FRAIL by Multidimensional Geriatric Assessment (MGA)
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
OS | 5 years
  Overall survival

SECONDARY OUTCOMES:
PFS | 5 years
  Progression free survival
FFS | 5 years
  Failure Free Survival
Response to initial therapy | 5 years
Early mortality rate | 5 years
% of patients who performed pre-phase therapy | 5 years
  Come to the prefect Therapy is a steroid-based therapy (administered at dosage of at least 25 mg / day) and / or vincristine, which precedes the beginning of the program of chemoimmunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spina, MD, Principal Investigator — CRO-Centro di Riferimento Oncologico
Locations (55):
- Italy (55):
  - Azienda Ospedaliera Caravaggio, Treviglio, Bergamo
  - A.O.Cardinale Panico Ematologia e centro trapianti, Tricase, LE
  - IRCCS Humanitas, Rozzano, Milano
  - CRO-Centro di Riferimento Oncologico, Aviano, Pordenone
  - CROB, Rionero in Vulture, Potenza
  - Polo Pontino, Latina, Roma
  - ASL TO-4, Ivrea, Torino
  - Ospedale S. Giacomo di Castelfranco Veneto, Castelfranco Veneto, Treviso
  - AO SS.Antonio e Biagio, Alessandria
  - AOU Ospedali Riuniti, Ancona
  - A.O. Universitaria Ospedale Consorziale Policlinico Di Bari, Bari
  - IRCC Istituto tumori Ematologia, Bari
  - AO Barletta, Barletta
  - SOS Ematologia Divisione Medicina Interna Ospedale degli Infermi, Biella
  - Spedali Civili di Brescia, Brescia
  - Ospedale Businco, Cagliari
  - Arnas Garibaldi, Catania
  - AO di Cosenza, Cosenza
  - AO Santa Croce e Carle, Cuneo
  - AOU Careggi, Florence
  - Ematologia Ospedale Vito Fazzi, Lecce
  - USL 6 Livorno Centro Aziendale Ematologia, Livorno
  - Ospedale di Matera, Matera
  - Area Vasta Romagna e IRST, Meldola (FC)
  - Ospedali Riuniti Papardo, Messina
  - Fondazione IRCCS Ca' Granda- Ospedale Maggiore Policlinico, Milan
  - Ospedale S. Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - AO Niguarda, Milan
  - Osp. San Carlo Borromeo Divisione di Oncologia Medica, Milan
  - AOU Policlinico di Modena, Modena
  - Ospedale San Gerardo, Monza
  - AUO Maggiore della Carità, Novara
  - Istituto Oncologico Veneto, Padua
  - AOU Padova, Padua
  - A.O. Universitaria Policlinico Giaccone Di Palermo, Palermo
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico S.Matteo, Pavia
  - AO di Perugia S. Maria della misericordia, Perugia
  - Ospedale di Pescara, Pescara
  - Ospedale Civile di Piacenza, Piacenza
  - Ospedale S. Maria delle Croci, Ravenna
  - A.O. Bianchi Melacrino Morelli, Reggio Calabria
  - AO Santa Maria Nuova, Reggio Emilia
  - Ospedale degli Infermi, Rimini
  - AOU La Sapienza, Roma
  - Policlinico Universitario A.Gemelli, Roma
  - Azienda OSpedaliera S. Andrea, Roma
  - AOU Senese, Siena
  - AO Santa Maria di Terni, Terni
  - AO Città della Salute e della Scienza Ematologia Universitaria, Torino
  - AO Città della Salute e della Scienza SC Ematologia, Torino
  - Ospedale di Circolo, Varese
  - Presidio Ospedaliero S. Andrea, Vercelli

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Merli F, Luminari S, Tucci A, Arcari A, Rigacci L, Hawkes E, Chiattone CS, Cavallo F, Cabras G, Alvarez I, Fabbri A, Re A, Puccini B, Barraclough A, Delamain MT, Ferrero S, Usai SV, Ferrari A, Cencini E, Pennese E, Zilioli VR, Marino D, Balzarotti M, Cox MC, Zanni M, Di Rocco A, Lleshi A, Botto B, Hohaus S, Merli M, Sartori R, Gini G, Nassi L, Musuraca G, Tani M, Bottelli C, Kovalchuk S, Re F, Flenghi L, Molinari A, Tarantini G, Chimienti E, Marcheselli L, Mammi C, Spina M. Simplified Geriatric Assessment in Older Patients With Diffuse Large B-Cell Lymphoma: The Prospective Elderly Project of the Fondazione Italiana Linfomi. J Clin Oncol. 2021 Apr 10;39(11):1214-1222. doi: 10.1200/JCO.20.02465. Epub 2021 Feb 12. PMID 33577377